CLINICAL TRIAL: NCT06017947
Title: Evaluation of a Musical Intervention on the Anxiety of Patients With a Diagnosis of Acute Coronary Syndrome in a Pre-Hospital Emergency Situation: MuSCA Randomized Controlled Trial
Acronym: MuSCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/CHU/02
Record Dates: First submitted 2023-03-16; First posted 2023-08-30 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard process (No Intervention)
- Musical intervention (Experimental)
  Interventions: Procedure: Music care

INTERVENTIONS:
Procedure: Music care — 20 min music listening during transportation to hospital
  Arms: Musical intervention

SUMMARY:
Acute coronary syndrome (ACS) encompasses a continuum of clinical situations secondary to acute myocardial ischemia. In France, it is a major health problem and represented 60,000 to 65,000 hospitalizations in 2010. In 2015, a diagnosis of ACS was made in 15 to 25% of patients consulting for chest pain in emergency medicine.

The incidence of ACS is estimated between 80,000 and 100,000 new cases per year. At the University Hospital Center (CHU) of Réunion, acute chest pain is the leading cause of discharges from the Mobile Emergency and Resuscitation Service (SMUR). In 2019, it represented 23% of exits, 8.5% of which concerned SCAs.

The SCA can be anxiety-provoking due to its unexpected and brutal nature. Pain related to myocardial ischemia generates anxiety. This increases when patients associate these pains with death. This anxiety is exacerbated by waiting times for care, especially for patients living in rural areas. In addition, conditions relating to medical care such as noise and the pre-hospital medical environment are perceived as influencing anxiety by patients.

The prevalence of anxiety is high, ranging from 30 to 48.5%, in patients with chest pain and/or ACS. A 2020 meta-analysis revealed that anxious patients at the start of their ACS treatment had an increased risk of death, non-fatal myocardial infarction, rehospitalization, recurrence of ACS and the need for coronary revascularization repeated. Overall, ACS patients with anxiety have a 21% increased risk of mortality and 47% increased risk of adverse cardiovascular events compared to those without anxiety.

Pre-hospital anxiolytic treatment is therefore essential and consists above all in reassuring the patient with ACS. Medicated anxiolytics are often combined with analgesics and recommended in front of a picture of agitation due to anxiety. However, negative effects may interfere, making clinical monitoring of these patients unsuitable. At the same time, several studies note that anxiety is underdiagnosed and undertreated in the care of these patients.

In reducing the anxiety of patients with ACS, unconventional care techniques such as aromatherapy or touch massage have demonstrated their effectiveness. Music therapy is recognized in reducing the anxiety of patients in intensive care or Cardiology.

To the knowledge, in France, the effect of a musical intervention on patients with pre-hospital ACS has not yet been studied. It is in this context that the MuSCA study takes place.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* With an established or suspected Acute Coronary Syndrome diagnosis
* With a stable clinical condition at the initial assessment:
* Whose anxiety assessment is > or = 30/100 mm on the Visual Analogue Scale
* Having provided express, free and informed consent
* With an estimated transport time of at least > 30 minutes

Exclusion Criteria:

* Under guardianship, curatorship or judicial safeguard procedure
* With hearing and visual impairments
* Participating in another clinical trial or having already been included in this study.
* Supported by helicopter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Anxiety change | 20 minutes
  This is to assess whether a 20-minute musical intervention associated with the usual care would reduce the anxiety of the patient suffering from an acute coronary syndrome in pre-hospital during his transfer to a health establishment. (intervention group) compared to usual management alone (control group).
  measurement méthod : analog visual scale

SECONDARY OUTCOMES:
Pain change | 20 minutes
  assess whether a musical intervention associated with the usual care allows a reduction, during the transfer to a health establishment of the pain score (Numerical Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Saint-Pierre, Île de La Réunion, France

IPD SHARING:
Plan to Share IPD: No